CLINICAL TRIAL: NCT04271865
Title: Dates a Food Treasure: Use of Dates Fruit in Alleviating and Managing Therapy-induced Anaemia for Hepatitis C Patients in Seven Villages of Egypt With Improving Their Quality of Life
Brief Title: Dates a Food Treasure in Alleviating Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Collaborators: Taibah University (Other); Rotary club of Heliopolis Sporting, Egypt (Unknown); Australian Embassy of Egypt (Unknown); Sustainable Development Project in the Kingdom of Saudi Arabia (KSA) (Unknown)
Responsible Party: Principal Investigator, Prof.Dr. Ammal Mokhtar Metwally, Principal Investigator, National Research Centre, Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20171226
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Anemia, Iron Deficiency
Keywords: HCV treated patients; Anemia; Dates
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia

STUDY DESIGN:
Intervention Model Description: providing Dates fruits as a potential palliative remedy to mitigate anaemia combined with nutritional education
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- therapy induced anemia for HCV treated patients (Other): Four types of interventions:
  * Educational to increase the number of nutritionally balanced meals and increase the frequency of iron-rich foods per day and improve current and risky nutritional habits
  * Provision of Dates : Dates fruit intake for all the anaemic patients
  * Recipe book
  * Model kitchen for all patients having Hemoglobin lower than normal hemoglobin levels; less than 13.2 grams (g) of hemoglobin per deciliter (dL) of blood for men and less than 11.6 for women.
  Interventions: Other: Nutritional Education; Other: model nutrition kitchen; Other: recipe book; Other: Provision of Dates

INTERVENTIONS:
Other: Nutritional Education — Provision of weekly awareness and educational sessions for 6 months. Sessions were conducted at the community based associations within the cases respective villages. Cases were subjected to 24 sessions for improving the patients' own nutrition situation through nutritional education about food rich in iron and counselling. The sessions focused on basic knowledge on iron deficiency anaemia, the most common presenting symptoms, iron rich dietary sources, factors that enhance and inhibit iron absorption, effects of anaemia on health and how to prevent it, Role of dates fruit in preventing and treating anaemia. Th e sessions also focused on the provision of a diverse range of local iron rich food. Special focus was on increasing patients' awareness for self-management of their status
Other: model nutrition kitchen — Implementing model nutrition kitchen; once every month for six months with six sessions for each village (6 sessions/village) with cooking sessions was done to promote eating healthy and provide innovative ideas for feeding anaemic cases. 117 patients were reached by the nutritional kitchen activities with 6 sessions until the end of the project. Special focus was done on skills like sharing cooking, meal planning, and label reading that help support healthy eating patterns. Suggesting ways that individuals can model healthy eating behaviors for friends and family members that is based on Dates fruit was encouraged.
Other: recipe book — 3) Development of recipe book that is based on the local food in the market to increase the number of nutritionally balanced meals and increase the frequency of iron-rich foods per day and improve current and risky nutritional habits
Other: Provision of Dates — Dates fruit intake for all the anaemic patients was provided for 16 weeks (four months):
  • Diagnosed anemic patients were given five to seven pieces of Dates (dependent on its weight) on daily basis for 16 weeks (each date fruits is about 10 -20 gm). Dates was taken as breakfast on daily base.
  The Dates fruit that was used during the proposed trial is Saudi's Dates extract know as Barni which is organic Dates. The fruit is mentioned more than 20 times in the Quran, This Barni is known for its very high nutritive value (vitamins, minerals and antioxidants) compared with other Dates types. The nutritive value of Barni is shown in the below table, calculated per every 100 gram (range 5- 10 pieces) of dry weight (DW) :
  The nutritive value of Barni calculated per every 100 gram (average 7-10 pieces) of dry weight (DW) of which iron constitutes 6.78 mg that represent 67.8 % of the recommended dietary allowance (RDA) of the males and 45.20 % of the RDA of the females

SUMMARY:
Introduction: In May 2016, seven villages in three governorates of Egypt were declared to be the first villages free from hepatitis C upon eliminating HCV virus by treatment with Sofosbuvir plus ribavirin (an interferon-free regimen). These patients were amounted to 2340 cases out of 19,991 screened residents of the seven villages within three governorates of Egypt. Although this combination was proved effective (95 %) in treatment of HCV genotype 4 among Egyptians, yet it resulted in anaemia with decreased quality of life for the majority of the treated HCV patients.

Aim of the project: To assess and manage therapy-induced anaemia among 2340 treated chronic hepatitis C patients with Sofosbuvir plus ribavirin, and improving their quality of life by provision of a comprehensive nutritional interventions that is based on Dates fruit intake.

Methodology: Dates fruit intake for all the diagnosed anaemic patients was provided for 16 weeks (four months). Five pieces of Dates fruit were taken as breakfast on daily basis (each date fruits is about 10 -20 gm). The Dates fruit that was used was Saudi's Dates extract known as Barni which is organic Dates. This Barni is known for its very high nutritive value (vitamins, minerals and antioxidants) compared with other Dates types. This Dates was imported from Saudi Arabia as donation through collaboration between NRC with Taibah University and Sustainable Development Project in the Kingdom of Saudi Arabia (KSA). In addition to Dates fruit intake, nutritional education to alleviate their anaemia was also provided. Haemoglobin level, risk of malnutrition and health-related quality of life (HRQoL) were assessed in all anemic patients before and after four months of intervention.

DETAILED DESCRIPTION:
Anaemia is a condition in which the number of red blood cells or their oxygen-carrying capacity is insufficient to meet physiologic needs. Anemia is a condition characterized by a decrease in the concentration of hemoglobin in the blood. Hemoglobin is necessary for transporting oxygen to tissues and organs in the body. Iron deficiency is thought to be the most common cause of anaemia globally. Iron deficiency anemia is due to insufficient iron that is necessary to produce enough red blood cells that enables them to carry oxygen (hemoglobin). As a result, iron deficiency anemia is associated with fatigue, general body weakness, frequent tiredness, dizziness and lowered resistance to disease and drowsiness. Overall, morbidity and mortality risks increase for individuals suffering from anemia, a condition in which blood lacks adequate healthy red blood cells. Red blood cells carry oxygen to the body's tissues.

Anemia is considered a serious public health problem worldwide with prevalence of 43% in the developing countries and of 9% in the developed ones. Research demonstrates that the majority of HCV treated patients with ribavirin became anaemic after treatment and they claimed that their quality of life was affected because of anaemia. Anaemia is one of the common side effects for Hepatitis C treated with ribavirin and remains a prominent concern. Partially, because Ribavirin destroys red blood cells by causing them to break open, or rupture and partially because of malnutrition due to the loss of appetite accompanying the treatment. Moreover addition of direct acting antiviral as Sofosbuvir to peginterferon plus ribavirin (PegIFN/RBV) increases the frequency as well as the severity, and hence, clinical relevance of anaemia, which has now become one of the major complications associated with hepatitis C therapy. Most significant factors associated with anaemia in patients receiving triple therapy include older age, lower body mass index (BMI), advanced fibrosis, and lower baseline haemoglobin.

Hemoglobin lower than normallevels indicate anemia; The normal hemoglobin range is generally defined as 13.2 to 16.6 grams (g) of hemoglobin per deciliter (dL) of blood for men and 11.6 to 15. g/dL for women. Severe anemia is manifested when Hb level is less than 8 grams (g) of hemoglobin per deciliter (dL) for both adult men aged 15 years and above and non- pregnant women aged 15 years and above Overall objective To help program planners plan regimens and guidelines to overcome therapy-induced anaemia with the use of functional food Objectives for direct beneficiaries

1. Improving the lives of the anaemic patients by providing a set of interventions for to alleviate their anaemia
2. improving participants' quality of life which was Dates fruits dependant.

This study was conducted as three phases:

The first phase included:

1. Equipping the three main primary health care units by automated cell counter
2. Training of the primary health care technicians to carry out screening for risk of anaemia
3. Screening and assessing incidence of anaemia and measuring haemoglobin concentration (Hb) among 2341 HCV treated cases (>18 years to 70 years) followed by confirming the anaemic status
4. Assessing the nutritional pattern and quality of life for the anaemic cases

The second phase included:

* Development of recipe book to increase the number of nutritionally balanced meals and increase the frequency of iron-rich foods per week
* Provision of awareness and educational sessions at the community based associations for improving the patients' own nutrition situation through nutritional education about food rich in iron and counselling. Special focus will be on increasing patients' awareness for self-management of their status.
* Provision of Dates : Dates fruit intake for all the anaemic patients was provided for 16 weeks (four months):Diagnosed anemic patients were given five pieces of Dates on daily basis for 16 weeks (each date fruits is about 10 -20 gm), of Dates. Dates was taken as breakfast on daily base.
* Provision of demonstration kitchen model

the third phase was the evaluation phase for :

1. Measuring change in the haemoglobin level
2. Measuring the change of the nutritional habits for all anaemic cases'
3. Measuring change of the quality of life indicators

Monitoring process:

A monthly monitoring sheet containing pictures and photos for the types of food was used for follow up of dietary habits. It was filled daily by the cases starting from the first day after the session for one month. Follow up was done for 6 months

ELIGIBILITY:
Inclusion Criteria:

* therapy induced anemia (HCV treated cases with anemia)

Hemoglobin lower than normal levels indicating mild and moderate anemia. The normal hemoglobin range is generally defined as 13.2 to 16.6 grams (g) of hemoglobin per deciliter (dL) of blood for men and 11.6 to 15. g/dL for women.

Exclusion Criteria:

* Severe anemia is manifested when HB level is less than 8 grams (g) of hemoglobin per deciliter (dL) for both adult men aged 15 years and above and non- pregnant women aged 15 years and above

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2017-02-26 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-12-25 (Actual)

PRIMARY OUTCOMES:
Percent change of the mean Hb level as a result of interventions | Four months after the initiation of the intervention
  The normal hemoglobin range is generally defined as 13.2 to 16.6 grams (g) of hemoglobin per deciliter (dL) of blood for men and 11.6 to 15. g/dL for women. This is according toWorld Health Organization (WHO) for the diagnosis of anaemia and assessment of severity.
  Screening for anaemia by Hemo-Cue then confirmation by the automated cell counter for assessing the incidence of anaemia and measuring haemoglobin concentration (Hb) Both serum iron and ferritin level were measured for confirming the severity of anaemia; mild, moderate and severe anaemia
percent change of the severity of anaemia | difference from the initial (before the intervention) with that four months after the initiation of the intervention
  The percent change of the severity of anaemia from mild to moderate or severe and the reversed was measured as per each participants

SECONDARY OUTCOMES:
Percent change of diet quality as a result of the interventions (as measured by the Diet Quality Index (DQI) | The difference from the initial (before the intervention) with that of four months after the initiation of the intervention
  The Diet Quality Index (DQI) is an instrument developed to measure overall diet quality that reflects a risk gradient for diet-related chronic disease. Dietary moderation and diversity are 2 new components. DQI-R scores range from 0 to 10 for each component, for a highest possible diet quality score of 100.
  Three levels of malnutrition were defined according to DQI :
  for the risk of anemia and malnutrition :At risk: below 40
  * Possible at risk: 40-50
  * Not at risk: more than 50
Percent change of the Health related quality of life (HRQoL) as a result of interventions | The difference from the initial (before the intervention) with that of four months after the initiation of the intervention
  SF-36 questionnaire for quality of life was implemented. The instrument is extensively validated and has been widely used for assessment of HRQoL in various settings including clinical trials . The questionnaire was provided in Arabic and this was done in the patients' villages. The SF-36 includes 36 questions about patients' perception of wellbeing, health status and daily functioning, which are used to calculate 8 HRQoL domain scores, each ranging from 0 to 100 with higher scores indicating better health: Physical Functioning (PF), Role Physical (RP), Bodily Pain (BP), General Health (GH), Vitality (VT), Social Functioning (SF), Role Emotional (RE), and Mental Health (MH).

CONTACTS AND LOCATIONS:
Overall Officials: Ammal M Metwally, Principal Investigator — National Research Centre, Egypt
Locations (1):
- National Research Centre, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) that underlie in a publication results will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after the study publication
Access Criteria: the data will be accessed through a link

REFERENCES:
- [Background] WHO. Haemoglobin concentrations for the diagnosis of anaemia and assessment of severity. Vitamin and Mineral Nutrition Information System. Geneva, World Health Organization, 2011 (WHO/NMH/NHD/MNM/11.1)
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Newby PK, Hu FB, Rimm EB, Smith-Warner SA, Feskanich D, Sampson L, Willett WC. Reproducibility and validity of the Diet Quality Index Revised as assessed by use of a food-frequency questionnaire. Am J Clin Nutr. 2003 Nov;78(5):941-9. doi: 10.1093/ajcn/78.5.941. PMID 14594780
- [Background] Rock W, Rosenblat M, Borochov-Neori H, Volkova N, Judeinstein S, Elias M, Aviram M. Effects of date ( Phoenix dactylifera L., Medjool or Hallawi Variety) consumption by healthy subjects on serum glucose and lipid levels and on serum oxidative status: a pilot study. J Agric Food Chem. 2009 Sep 9;57(17):8010-7. doi: 10.1021/jf901559a. PMID 19681613
- [Background] Al-Radadi, N.S. Green synthesis of platinum nanoparticles using Saudi's Dates extract and their usage on the cancer cell treatment. Arabian Journal of Chemistry .2019; 12, 330-349